CLINICAL TRIAL: NCT01368107
Title: A Randomised, Multicentric, Phase 2a Study Evaluating the Impact of an Immunotherapy by IL-7 on CD4 Lymphopenia, Risks of Severe Haematological Toxicity and Tumor Progression in Metastatic Breast Cancer Patients
Brief Title: Study Evaluating Impact of IL-7 on CD4 Lymphopenia, Risks of Severe Haematological Toxicity and Tumor Progression in Metastatic Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Ministry of Health, France (Other Government); Cytheris, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELYPSE 7; 2011-000226-30 (EudraCT Number)
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2013-12

CONDITIONS: Metastatic Breast Cancer
Keywords: IL-7; metastatic breast cancer patients; lymphopenia
MeSH Terms: conditions — Breast Neoplasms; Lymphopenia | interventions — Interleukin-7

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo Arm (Placebo Comparator): the patients will receive Placebo before the 1st and during the 3rd CT cycle (N=6)
  Interventions: Drug: placebo
- CYT107 treatment before CT (Experimental): patients will receive an induction cycle of CYT107 (10µg/kg/week subcutaneously for 3 weeks) before the 1st CT cycle and the placebo during the 3rd CT cycle (N=6)
  Interventions: Drug: placebo; Drug: interleukin 7
- CYT107 treatment during CT (Experimental): patients will receive the placebo before the 1st CT cycle and a delayed treatment with CYT107 (10µg/kg/week subcutaneously for 3 weeks) during the 3rd CT cycle (N=6)
  Interventions: Drug: interleukin 7
- CYT107 treatment before and during CT (Experimental): patients will receive an induction cycle of CYT107 (10µg/kg/week subcutaneously for 3 weeks) before the 1st CT cycle and a maintenance cycle of IL-7 (10µg/kg/week subcutaneously for 3 weeks) during the 3rd CT cycle (N=6).
  Interventions: Drug: interleukin 7

INTERVENTIONS:
Drug: placebo — Placebo before the 1st (D0, D7, D14)and during the 3rd CT cycle (D57, D64, D71)
  Arms: CYT107 treatment before CT; Placebo Arm
Drug: interleukin 7 — patients will receive an induction cycle of CYT107 (10µg/kg/week subcutaneously for 3 weeks) before the 1st CT cycle (D0, D7, D14) and the placebo during the 3rd CT cycle (D57, D64, D71)
  Arms: CYT107 treatment before CT
Drug: interleukin 7 — patients will receive the placebo before the 1st CT cycle (D0, D7, D14) and a delayed treatment with CYT107 (10µg/kg/week subcutaneously for 3 weeks) during the 3rd CT cycle (D57, D64, D71)
  Arms: CYT107 treatment during CT
Drug: interleukin 7 — patients will receive an induction cycle of CYT107 (10µg/kg/week subcutaneously for 3 weeks) before the 1st CT cycle (D0, D7, D14) and a maintenance cycle of IL-7 (10µg/kg/week subcutaneously for 3 weeks) during the 3rd CT cycle (D57, D64, D71)
  Arms: CYT107 treatment before and during CT

SUMMARY:
The purpose of the study is to evaluate the impact of an immunotherapy by IL-7 on CD4 lymphopenia, risks of severe haematological toxicity and tumor progression in metastatic breast cancer patients.

The primary objective is to determine the optimal schedule to deliver CYT107 during chemotherapy based on restoration of CD4 count.

This study is a phase II, randomised, double-blind, placebo-controlled, single-centre.

24 patients will be included in the study.

DETAILED DESCRIPTION:
A key secondary objective is to determine if CYT107 treatment enables to reduce the incidence of severe haematological toxicity (any type of haematological toxicity Grade ≥ 3) post-chemotherapy.

Other secondary objectives are to assess the impact of CYT107 treatment on the following parameters:

* Overall incidence of side effects (any type any grade)
* Progression-free survival (PFS)
* Compliance to chemotherapy regimen (dose intensity, number of chemotherapy cycles).
* CD4 lymphopenia over the study period

Exploratory biological markers

A series of biomarkers analyses will be performed to evaluate if CYT107 treatment will:

* selectively stimulate the proliferation and activation of peripheral immune subsets (analysis of phenotype and activation status of peripheral immune e sub-populations)
* selectively improve the functional response of T cells, DC subsets and NK cells.
* is able to revert tolerogenic immune burden to increase specific anti-tumor response (measure of antigen specific CD8 response, measure of cytokine plasmatic levels)
* enable to increase TCR diversity (analysis of combinatorial diversity).

ELIGIBILITY:
Inclusion Criteria:

* Female aged more than 18 years
* Histologic diagnosis of metastatic breast cancer to be treated with capecitabine at study entry. NB: Patients previously treated with capecitabine are eligible only if more than 6 months have elapsed since the last capecitabine intake.
* Lymphopenic (i.e. with at least one value of lymphocyte count 1500/µL within 15 days before Day 0).
* Performance status ECOG of 0, 1,2 or 3
* Life expectancy ≥ 6months
* Adequate bone marrow, hepatic and renal function as follows:

  * Neutrophils ≥ 1,000/µL
  * Platelets ≥ 100 109/µL
  * ASAT, ALAT, or Alkaline Phosphatase ≤ 2.5 x ULN
  * Total Bilirubin ≤ 1.5 x ULN
  * INR ≤ 1.5
  * Calculated creatinin clearance ≥ 60mL/min (Cockcroft formula or MDRD formula for patients older than 65 years old)- Ability to understand and sign informed consent
* Covered by a medical insurance.

Exclusion Criteria:

* Prior history of other malignancies other than breast cancer (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) unless the subjects has been free of the disease for at least 3 years.
* No resolution of specific toxicities related to any prior anti-cancer therapy to Grade ≤2 according to the NCI CTCAE v.4.0 (except lymphopenia, alopecia and neuropathy)
* Wash out period of less than 5 times the half-life of previous anti-cancer treatment before study entry, except if previous chemotherapy treatment before study entry. NB: For patient previously treated by hormonotherapy, a wash out period of 1 week will be sufficient
* Uncontrolled hypertension (i.e., resting systolic blood pressure greater than140 mmHg or resting diastolic blood pressure greater than 90 mmHg), despite pharmacologic antihypertensive treatment, confirmed with a second blood pressure measurement done later in the same day
* History of lymphoid malignancy (e.g. Hodgkin disease, non Hodgkin lymphoma, Leukemia).
* History of splenectomy or hematologic disease associated with hypersplenism, such as gamma or beta-thalassemia, hereditary spherocytosis, Gaucher's disease, or autoimmune hemolytic anemia.
* Any cardiac, pulmonary, thyroid, renal, hepatic, neurological severe/uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol
* Any history of severe auto-immune disease
* Hepatitis B antigen (HBs Ag) positive, Hepatitis C (HCV Ab) antibody positive or HCV RNA detectable
* Documented HIV-1 positivity
* History of cardiovascular disorders grade >2 (NYHA) within 6 months preceding the inclusion
* Active uncontrolled viral, fungal or bacterial infection
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements (participants must agree to refrain from substance abuse use during the entire course of the study)
* Pregnant or breast-feeding women
* No use of effective birth control methods for women of childbearing potential
* Any contraindications to capecitabine treatment (refer to Xeloda SPC Appendix 11) and to any other anti-cancer treatment authorized as per protocol (refer to respective SPC for specific contraindications)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
to determine the optimal schedule to deliver CYT107 during chemotherapy based on restoration of CD4 count | after 11 weeks of treatment
  Evolution of CD4 count from Day 0 to Week 11 with repeated measures from D0 to W12 (D0, D21, D57, D78).

SECONDARY OUTCOMES:
to determine if CYT107 treatment enables to reduce the incidence of severe haematological toxicity (any type of haematological toxicity Grade ≥ 3) post-chemotherapy | at the end of study M12
To assess the impact of CYT107 on progression-free survival | at the end of study (M12)
  Time from randomisation to first evidence of progression or death of any cause.
To assess the impact of CYT107 on compliance to chemotherapy regimen (dose intensity, number of chemotherapy cycles). | at the end of study (M12)
  Number of CT cycles, CT dose delays and/or reduction, CT discontinuation
To assess the impact of CYT107 on CD4 lymphopenia over the study period | at the end of study (M12)
  Evolution of CD4 count from Day 0 to end of study visit
to evaluate if CYT107 treatment will selectively stimulate the proliferation and activation of peripheral immune subsets (analysis of phenotype and activation status of peripheral immune e sub-populations) | D0, D21, D57, D78 and at end of study M12
  Measure of frequency and activation status of circulating immune subpopulations on fresh whole blood. Multi-parametric marker sets (6-8 markers) will be used to analyse phenotype of immune subpopulations (TCD4+, TCD8+, Treg, T, NK, DC) and their activation status (PD1, ICOS, CD39, CD73, CD62L, CCR7, CD45RO, CD45RA, CD86).
to evaluate if CYT107 treatment will selectively improve the functional response of T cells, DC subsets and NK cells | D0, D21, D57, D78 and at the end of study M12
  Analysis of the functional response of T cells, DC subsets and NK cells
to evaluate if CYT107 treatment will is able to revert tolerogenic immune burden to increase specific anti-tumor response (measure of antigen specific CD8 response, measure of cytokine plasmatic levels) | D0, D21, D57, D78 and at the end of study M12
  * Analysis of tumor associated antigen (TAA) specific CD8 responses
  * Quantification of circulating cytokines including mainly, but not limited to, IL-6, IL-2, IFN, VEGF, TNF, IL-15,F FGF using Luminex technology and VEGF, TGF, IL-7R by Elisa.
to evaluate if CYT107 treatment will enable to increase TCR diversity (analysis of combinatorial diversity). | D0, D21, D57, D78 and at the end of study M12
  Evaluation of T cell receptor diversity using ImmuneTraCkeR test and Constel'ID software (ImmunID Technologies, Grenoble, France).
To assess the impact of CYT107 treatment on overall incidence of side effects | after 12 weeks of treatment
  Number of patients with AEs (any type any grade) using NCI-CTCAE scale (version 4.0) from D0 to W12

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Ray Coquart, Principal Investigator — Centre Léon Bérard, Lyon
Locations (3):
- France (3):
  - Centre Leon Berard, Lyon
  - Institut Curie, Paris
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Zou W. Regulatory T cells, tumour immunity and immunotherapy. Nat Rev Immunol. 2006 Apr;6(4):295-307. doi: 10.1038/nri1806. PMID 16557261
- [Result] Treilleux I, Blay JY, Bendriss-Vermare N, Ray-Coquard I, Bachelot T, Guastalla JP, Bremond A, Goddard S, Pin JJ, Barthelemy-Dubois C, Lebecque S. Dendritic cell infiltration and prognosis of early stage breast cancer. Clin Cancer Res. 2004 Nov 15;10(22):7466-74. doi: 10.1158/1078-0432.CCR-04-0684. PMID 15569976
- [Result] Bates GJ, Fox SB, Han C, Leek RD, Garcia JF, Harris AL, Banham AH. Quantification of regulatory T cells enables the identification of high-risk breast cancer patients and those at risk of late relapse. J Clin Oncol. 2006 Dec 1;24(34):5373-80. doi: 10.1200/JCO.2006.05.9584. PMID 17135638
- [Result] Gobert M, Treilleux I, Bendriss-Vermare N, Bachelot T, Goddard-Leon S, Arfi V, Biota C, Doffin AC, Durand I, Olive D, Perez S, Pasqual N, Faure C, Ray-Coquard I, Puisieux A, Caux C, Blay JY, Menetrier-Caux C. Regulatory T cells recruited through CCL22/CCR4 are selectively activated in lymphoid infiltrates surrounding primary breast tumors and lead to an adverse clinical outcome. Cancer Res. 2009 Mar 1;69(5):2000-9. doi: 10.1158/0008-5472.CAN-08-2360. Epub 2009 Feb 24. PMID 19244125
- [Result] Blay JY, Chauvin F, Le Cesne A, Anglaret B, Bouhour D, Lasset C, Freyer G, Philip T, Biron P. Early lymphopenia after cytotoxic chemotherapy as a risk factor for febrile neutropenia. J Clin Oncol. 1996 Feb;14(2):636-43. doi: 10.1200/JCO.1996.14.2.636. PMID 8636781
- [Result] Blay JY, Le Cesne A, Mermet C, Maugard C, Ravaud A, Chevreau C, Sebban C, Guastalla J, Biron P, Ray-Coquard I. A risk model for thrombocytopenia requiring platelet transfusion after cytotoxic chemotherapy. Blood. 1998 Jul 15;92(2):405-10. PMID 9657738
- [Result] Ray-Coquard I, Le Cesne A, Rubio MT, Mermet J, Maugard C, Ravaud A, Chevreau C, Sebban C, Bachelot T, Biron P, Blay JY. Risk model for severe anemia requiring red blood cell transfusion after cytotoxic conventional chemotherapy regimens. The Elypse 1 Study Group. J Clin Oncol. 1999 Sep;17(9):2840-6. doi: 10.1200/JCO.1999.17.9.2840. PMID 10561360
- [Result] Ray-Coquard I, Borg C, Bachelot T, Sebban C, Philip I, Clapisson G, Le Cesne A, Biron P, Chauvin F, Blay JY; ELYPSE study group. Baseline and early lymphopenia predict for the risk of febrile neutropenia after chemotherapy. Br J Cancer. 2003 Jan 27;88(2):181-6. doi: 10.1038/sj.bjc.6600724. PMID 12610500
- [Result] Marec-Berard P, Blay JY, Schell M, Buclon M, Demaret C, Ray-Coquard I. Risk model predictive of severe anemia requiring RBC transfusion after chemotherapy in pediatric solid tumor patients. J Clin Oncol. 2003 Nov 15;21(22):4235-8. doi: 10.1200/JCO.2003.09.121. PMID 14615453
- [Result] Borg C, Ray-Coquard I, Philip I, Clapisson G, Bendriss-Vermare N, Menetrier-Caux C, Sebban C, Biron P, Blay JY. CD4 lymphopenia as a risk factor for febrile neutropenia and early death after cytotoxic chemotherapy in adult patients with cancer. Cancer. 2004 Dec 1;101(11):2675-80. doi: 10.1002/cncr.20688. PMID 15503313
- [Result] Ray-Coquard I, Cropet C, Van Glabbeke M, Sebban C, Le Cesne A, Judson I, Tredan O, Verweij J, Biron P, Labidi I, Guastalla JP, Bachelot T, Perol D, Chabaud S, Hogendoorn PC, Cassier P, Dufresne A, Blay JY; European Organization for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group. Lymphopenia as a prognostic factor for overall survival in advanced carcinomas, sarcomas, and lymphomas. Cancer Res. 2009 Jul 1;69(13):5383-91. doi: 10.1158/0008-5472.CAN-08-3845. Epub 2009 Jun 23. PMID 19549917
- [Result] Fry TJ, Mackall CL. The many faces of IL-7: from lymphopoiesis to peripheral T cell maintenance. J Immunol. 2005 Jun 1;174(11):6571-6. doi: 10.4049/jimmunol.174.11.6571. PMID 15905493
- [Result] Menetrier-Caux C, Gobert M, Caux C. Differences in tumor regulatory T-cell localization and activation status impact patient outcome. Cancer Res. 2009 Oct 15;69(20):7895-8. doi: 10.1158/0008-5472.CAN-09-1642. Epub 2009 Oct 6. PMID 19808962
- [Result] Fry TJ, Moniuszko M, Creekmore S, Donohue SJ, Douek DC, Giardina S, Hecht TT, Hill BJ, Komschlies K, Tomaszewski J, Franchini G, Mackall CL. IL-7 therapy dramatically alters peripheral T-cell homeostasis in normal and SIV-infected nonhuman primates. Blood. 2003 Mar 15;101(6):2294-9. doi: 10.1182/blood-2002-07-2297. Epub 2002 Oct 31. PMID 12411295
- [Result] Fry TJ, Mackall CL. Interleukin-7: from bench to clinic. Blood. 2002 Jun 1;99(11):3892-904. doi: 10.1182/blood.v99.11.3892. No abstract available. PMID 12010786
- [Result] Rosenberg SA, Sportes C, Ahmadzadeh M, Fry TJ, Ngo LT, Schwarz SL, Stetler-Stevenson M, Morton KE, Mavroukakis SA, Morre M, Buffet R, Mackall CL, Gress RE. IL-7 administration to humans leads to expansion of CD8+ and CD4+ cells but a relative decrease of CD4+ T-regulatory cells. J Immunother. 2006 May-Jun;29(3):313-9. doi: 10.1097/01.cji.0000210386.55951.c2. PMID 16699374
- [Result] Sportes C, Hakim FT, Memon SA, Zhang H, Chua KS, Brown MR, Fleisher TA, Krumlauf MC, Babb RR, Chow CK, Fry TJ, Engels J, Buffet R, Morre M, Amato RJ, Venzon DJ, Korngold R, Pecora A, Gress RE, Mackall CL. Administration of rhIL-7 in humans increases in vivo TCR repertoire diversity by preferential expansion of naive T cell subsets. J Exp Med. 2008 Jul 7;205(7):1701-14. doi: 10.1084/jem.20071681. Epub 2008 Jun 23. PMID 18573906
- [Result] Akashi K, Kondo M, von Freeden-Jeffry U, Murray R, Weissman IL. Bcl-2 rescues T lymphopoiesis in interleukin-7 receptor-deficient mice. Cell. 1997 Jun 27;89(7):1033-41. doi: 10.1016/s0092-8674(00)80291-3. PMID 9215626
- [Result] Li WQ, Guszczynski T, Hixon JA, Durum SK. Interleukin-7 regulates Bim proapoptotic activity in peripheral T-cell survival. Mol Cell Biol. 2010 Feb;30(3):590-600. doi: 10.1128/MCB.01006-09. Epub 2009 Nov 23. PMID 19933849
- [Result] McFarland RD, Douek DC, Koup RA, Picker LJ. Identification of a human recent thymic emigrant phenotype. Proc Natl Acad Sci U S A. 2000 Apr 11;97(8):4215-20. doi: 10.1073/pnas.070061597. PMID 10737767
- [Result] Alpdogan O, van den Brink MR. IL-7 and IL-15: therapeutic cytokines for immunodeficiency. Trends Immunol. 2005 Jan;26(1):56-64. doi: 10.1016/j.it.2004.11.002. PMID 15629410
- [Result] Melchionda F, Fry TJ, Milliron MJ, McKirdy MA, Tagaya Y, Mackall CL. Adjuvant IL-7 or IL-15 overcomes immunodominance and improves survival of the CD8+ memory cell pool. J Clin Invest. 2005 May;115(5):1177-87. doi: 10.1172/JCI23134. Epub 2005 Apr 7. PMID 15841203
- [Result] Jaleco S, Swainson L, Dardalhon V, Burjanadze M, Kinet S, Taylor N. Homeostasis of naive and memory CD4+ T cells: IL-2 and IL-7 differentially regulate the balance between proliferation and Fas-mediated apoptosis. J Immunol. 2003 Jul 1;171(1):61-8. doi: 10.4049/jimmunol.171.1.61. PMID 12816983
- [Result] Sereti I, Dunham RM, Spritzler J, Aga E, Proschan MA, Medvik K, Battaglia CA, Landay AL, Pahwa S, Fischl MA, Asmuth DM, Tenorio AR, Altman JD, Fox L, Moir S, Malaspina A, Morre M, Buffet R, Silvestri G, Lederman MM; ACTG 5214 Study Team. IL-7 administration drives T cell-cycle entry and expansion in HIV-1 infection. Blood. 2009 Jun 18;113(25):6304-14. doi: 10.1182/blood-2008-10-186601. Epub 2009 Apr 20. PMID 19380868
- [Result] Levy Y, Lacabaratz C, Weiss L, Viard JP, Goujard C, Lelievre JD, Boue F, Molina JM, Rouzioux C, Avettand-Fenoel V, Croughs T, Beq S, Thiebaut R, Chene G, Morre M, Delfraissy JF. Enhanced T cell recovery in HIV-1-infected adults through IL-7 treatment. J Clin Invest. 2009 Apr;119(4):997-1007. doi: 10.1172/JCI38052. Epub 2009 Mar 16. PMID 19287090
- [Result] 26. Levy, Y., et al. Effects of r-hIL-7 on T-cell Recovery and Thymic Output in HIV-infected Patients receiving antiretroviral therapy (ART). Interim Analysis of a Phase I/IIa Multicenter Study. in ICAAC. 2009. San Francisco.
- [Result] 27. Miguel-Angel Perales, Jenna D. Goldberg,, Leuren Lechner Jianda Yuan, Esperanza Papadopoulos, James W. Young, Ann A. Jakubowski, Guenther Koehne, Humilidad Gallardo, Ryan Kendle, Cailian Liu, Teresa Rasalan, Yinyan Xu, Bushra Zaidi, Jedd D Wolchok, Therese Croughs, Michel Morre, Molly Maloy, Glenn Heller and Marcel R.M. van den Brink. Recombinant Human Interleukin-7 (CYT107) Enhances CD4 and CD8 T Cell Recovery Following T-Cell Depleted Allogeneic Hematopoietic Stem Cell Transplant In Patients with Myeloid Malignancies Oral and Poster Abstracts Oral Session: ASH 2010 Meeting.
- [Result] Li B, VanRoey MJ, Jooss K. Recombinant IL-7 enhances the potency of GM-CSF-secreting tumor cell immunotherapy. Clin Immunol. 2007 May;123(2):155-65. doi: 10.1016/j.clim.2007.01.002. Epub 2007 Feb 22. PMID 17320482
- [Result] Pellegrini M, Calzascia T, Elford AR, Shahinian A, Lin AE, Dissanayake D, Dhanji S, Nguyen LT, Gronski MA, Morre M, Assouline B, Lahl K, Sparwasser T, Ohashi PS, Mak TW. Adjuvant IL-7 antagonizes multiple cellular and molecular inhibitory networks to enhance immunotherapies. Nat Med. 2009 May;15(5):528-36. doi: 10.1038/nm.1953. Epub 2009 Apr 26. PMID 19396174
- [Result] McAlister FA, Straus SE, Sackett DL, Altman DG. Analysis and reporting of factorial trials: a systematic review. JAMA. 2003 May 21;289(19):2545-53. doi: 10.1001/jama.289.19.2545. PMID 12759326